CLINICAL TRIAL: NCT01063244
Title: Comparison of Foley Balloon With or Without Traction for the Cervical Ripening
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: St. Luke's Hospital, Pennsylvania (Other)
Responsible Party: Principal Investigator, James Anasti, MD, Director, OB?GYN Residency Program, St. Luke's Hospital, Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SLHN-08-21
Record Dates: First submitted 2010-02-03; First posted 2010-02-05 (Estimated); Last update posted 2016-04-18 (Estimated); Status verified 2016-04

CONDITIONS: Pregnancy
Keywords: pregnancy; induction of Labor; Cervical ripening; Foley balloon

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FoleyBalloon (Active Comparator): foley balloon placed in the cervix
  Interventions: Device: foley balloon only
- foley balloon with weight (Active Comparator): foley balloon with weight attached
  Interventions: Device: foley balloon with weight attached

INTERVENTIONS:
Device: foley balloon only — place foley balloon only in cervix
  Arms: FoleyBalloon
Device: foley balloon with weight attached — foley balloon with 1000cc IV bag attached
  Arms: foley balloon with weight

SUMMARY:
We will compare the use of foley bulb catheters placed in the cervix for ripening of the cervix for labor induction,.

DETAILED DESCRIPTION:
One arm will have the foley balloon placed alone in the cervix. And one arm will have the foley balloon placed in the cervix and then attached to a weight (1000 cc Iv Bag of fluid). Our hypothesis is that the weighted balloon will be more effective than the non-weighted balloon in the ripening of the cervix for induction of labor

ELIGIBILITY:
Inclusion Criteria:

* Term pregnancy scheduled for induction of labor

Exclusion Criteria:

* Preterm pregnancy that require induction for fetal indications

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2009-01; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Time to effectively ripen cervix | to effective cervical ripening

CONTACTS AND LOCATIONS:
Overall Officials: James N Aansti, MD, Principal Investigator — St. Luke's Hospital
Locations (1):
- St Luke's Hosptial & Health Network, Bethlehem, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No